CLINICAL TRIAL: NCT06642285
Title: Effect of Implementing Evidence Based Practices on Prevention of Associated Nasal Pressure Injuries Among Preterm Neonates With Non-Invasive Respiratory Support
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Kafrelsheikh University (Other)
Responsible Party: Principal Investigator, Eman Wardany Abdelaal Mohamed, assistant professor of pediatric nursing, Kafrelsheikh University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: KafrelsheikhU4
Record Dates: First submitted 2024-10-09; First posted 2024-10-15 (Actual); Last update posted 2024-10-15 (Actual); Status verified 2024-10

CONDITIONS: Mechanical Ventilation Complication; Respiratory Distress Syndrome in Premature Infant

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control Group (No Intervention): : it will include thirty premature neonates who will receive the usual hospital care in accordance with hospital protocols, without any extra procedures or therapies.
- Bundle group (Experimental): : it will include thirty premature neonates who will receive evidence-based guidelines on the prevention of nasal pressure injuries in form of a care bundle from the first day of providing NIRS till weaning.
  Interventions: Procedure: Non Invasive Respiratory Support bundle

INTERVENTIONS:
Procedure: Non Invasive Respiratory Support bundle — premature neonates who will receive evidence-based guidelines for prevention of nasal pressure injuries associated with non invasive respiratory support till weaning
  Arms: Bundle group

SUMMARY:
This study aims to evaluate the effect of implementing evidence based practices on prevention of associated nasal pressure injuries among preterm neonates with non invasive respiratory support

DETAILED DESCRIPTION:
The researchers explained the study's aim, benefits, and procedures for participation, after that the parents of the neonates provided an informed consent. Over a one-week period, staff education programs regarding Evidence-Based Guidelines for non-invasive respiratory support will be conducted for NICU nursing staff. These sessions, lasting 15 to 20 minutes, will be held during regularly scheduled work hours, with four different sessions will offer throughout the day. The preterm neonates' characteristics and clinical data will be extracted from their hospital records for the two groups on the first day of admission for both groups prior to intervention to identify those who fulfilled the current study's inclusion criteria. Neonatal baseline data was collected from their records on the first day of admission for the two groups prior to intervention in order to identify neonates who meet the required criteria of the study. Then the participants were selected and divided randomly (using a simple random method) into two equal groups. One subject for the control group, one for the study group and so on, distributed the participants into two equivalent groups as fellow:

Control Group: Consisted of 30 premature neonates who will receive conventional hospital care with no additional interventions.

Study Group: Consisted of 30 premature neonates who will receive 6 evidence-based practices on the prevention of nasal pressure injuries as follows:

* Use an appropriately sized nasal interface device.
* The Use of Skin Barrier Products between nasal skin and nasal interface device
* Visually examining the preterm newborn every hour to ensure appropriate nasal interface position
* Once every 12-hour shift, the protective barrier and nasal device are briefly removed to allow for a full nasal skin examination
* Follow developmental care principles by repositioning the infant every three to four hours.
* Pain scores should be taken at least every three to four hours.

ELIGIBILITY:
Inclusion Criteria:

* Preterm neonates receiving NIRS
* whose gestational ages ranges between 30 and 37 weeks, and both genders

Exclusion Criteria:

* all preterm neonates not receiving NIRS,
* have prior nasal trauma caused by tracheal intubation
* or Infants exhibiting evidence of nasal damage during the NIRS procedure,
* have upper respiratory abnormalities.
* preterm neonates who have undergone any type of surgery and had life-threatening congenital abnormalities.

Ages: 30 Weeks to 37 Weeks | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 30 (Estimated)
Dates: Start 2024-08-01 (Actual); Primary Completion 2024-12-30 (Estimated); Study Completion 2025-01-30 (Estimated)

PRIMARY OUTCOMES:
change from the baseline nasal skin integrity on Nasal injury classification tool | Researchers will assess the nasal skin of preterm infants every 3-6 hours from the first day of providing NIRS till 14 days to determine the nasal damage score in both groups.
  : it is adopted from (Fischer et al., 2010) based on the standardized classification of the decubitus lesions from the US National Pressure Ulcer Advisory Panel (NPUAP) (Black et al., 2007; The National Pressure Ulcer Advisory Panel, 1989). This tool will be employed to describe and track the progression and severity of nasal injuries caused by NIRS in neonates by assessing nasal region (the nasal tip, nasal septum, nostril, and nose shape change) for erythema, ulceration, and necrosis, in order to ensure proper and early treatment
change from the baseline pain score on Premature Infant Pain Profile (PIPP) | - Researchers will evaluate pain scores for preterm infants in both groups every 3-4 hours from the first day of providing NIRS till 14 days
  It will be adopted from (Stevens et al., 1996). The Premature Infant Pain Profile (PIPP) is a biobehavioral observational technique used to quantify acute and procedure pain in premature infants. It assesses seven indicators: gestational age, behavioral state, increased heart rate, decreased oxygen saturation, forehead bulging, eye squeezing, and nasolabial furrows. Each indicator is scored on a four-point Likert scale, from 0 to 3. The total PIPP score, which is the sum of points for all seven indications, varies between 0 to 21. Higher scores imply more painful conduct. A number of 0-6 indicates no pain, 7-12 indicates mild to moderate pain, and a score more than 12 indicates severe pain.

CONTACTS AND LOCATIONS:
Overall Officials: Eman W Wardany, ass. professor, Principal Investigator — pediatric nursing department, faculty of nursing kafrelsheikh univeristy
Locations (1):
- Kafrelsheikh University, Kafr ash Shaykh, Kafr el-Sheikh Governorate, Egypt

IPD SHARING:
Plan to Share IPD: No